CLINICAL TRIAL: NCT06996080
Title: A Randomized, Double-masked, Sham-controlled, Multicenter, Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal Tabirafusp Alfa (KSI-101) in Participants With Macular Edema Secondary to Inflammation (MESI) - PINNACLE
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal KSI-101 in Participants With Macular Edema Secondary to Inflammation (MESI) - PINNACLE
Acronym: PINNACLE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kodiak Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KSMP001-S2
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Macular Edema Secondary to Inflammation
Keywords: MESI; macular edema; inflammatory macular edema; macular edema associated with inflammation
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KSI-101 5 mg (Experimental): Intravitreal injection of KSI-101 5 mg once every 4 weeks for 6 monthly doses followed by individualized dosing
  Interventions: Drug: KSI-101
- KSI-101 10 mg (Experimental): Intravitreal injection of KSI-101 10 mg once every 4 weeks for 6 monthly doses followed by individualized dosing
  Interventions: Drug: KSI-101
- Sham (Sham Comparator): Sham injection once every 4 weeks for 6 monthly doses followed by individualized sham dosing
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Drug: KSI-101 — Intravitreal injection
  Other Names: tabirafusp alfa
  Arms: KSI-101 10 mg; KSI-101 5 mg
Other: Sham Comparator — Sham injections
  Arms: Sham

SUMMARY:
A Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal KSI-101 in Participants with Macular Edema Secondary to Inflammation (MESI)

ELIGIBILITY:
Inclusion Criteria:

* Patients with MESI, with a CST of ≥320 and <400 microns on SD-OCT and a BCVA score of ≥25 and ≤78 ETDRS letters (between ~20/25 and 20/320 Snellen equivalent) in the Study Eye at Day 1;
* Diagnosis of active or inactive non-infectious intraocular inflammation, acute or chronic in the Study Eye.

Exclusion Criteria:

* ME in the Study Eye secondary to diabetes, RVO, or wAMD
* Active or suspected ocular or periocular infection in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Mean change in BCVA | Week 24
  Mean change in BCVA from Day 1 to the average of Week 20 and Week 24.

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Research Network Arizona, Scottsdale, Arizona
  - Global Research Management, Inc., Glendale, California
  - UCLA Stein Eye Institute, Los Angeles, California
  - Stanford Byers Eye Institute, Palo Alto, California
  - California Eye Specialists Medical Group, Inc., Pasadena, California
  - California Eye Specialists Medical Group, Inc., Redlands, California
  - Retina Consultants of Southern California, Redlands, California
  - Retinal Consultants Medical Group Inc, Sacramento, California
  - Retina Group of New England, PC, Waterford, Connecticut
  - Retina Group of Florida (Ft. Lauderdale), Fort Lauderdale, Florida
  - Associated Vitreoretinal and Uveitis Consultants LLC, Carmel, Indiana
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Retina Consultants of Minnesota, Saint Louis Park, Minnesota
  - The Retina Institute, St Louis, Missouri
  - Retina Associates of New York, P.C., New York, New York
  - North Carolina Retina Associates (Cary), Cary, North Carolina
  - North Carolina Retina Associates (Wake Forest), Wake Forest, North Carolina
  - Cascade Medical Research Institute, Springfield, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Charleston Neuroscience Institute, LLC (Charleston), Charleston, South Carolina
  - Palmetto Retina Center (West Columbia), West Columbia, South Carolina
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Austin Retina Associates, PLLC (Austin), Austin, Texas
  - UT Austin, Austin, Texas
  - Retina Consultants of Texas (Bellaire), Bellaire, Texas
  - Texas Retina Center, Houston, Texas
  - Retina Consultants of Texas (Katy), Katy, Texas
  - Texas Retina Associates (Plano), Plano, Texas
  - Austin Retina Associates, PLLC (Round Rock), Round Rock, Texas
  - Retina Consultants of Texas (San Antonio), San Antonio, Texas
  - Retina Consultants of Texas (Woodlands), The Woodlands, Texas
  - Pacific Northwest Retina (Bellevue), Bellevue, Washington
  - Pacific Northwest Retina (Silverdale), Silverdale, Washington

IPD SHARING:
Plan to Share IPD: No